CLINICAL TRIAL: NCT02174588
Title: Moderate Sedation for Elective Upper Endoscopy With Balanced Propofol Versus Propofol Alone: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2012-0801
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: EGD Procedure
Keywords: sedation, propofol, midazolam
MeSH Terms: interventions — Midazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- balanced propofol group (Experimental)
  Interventions: Drug: Midazolam + propofol
- propofol alone group (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Midazolam + propofol — Midazolam and propofol are used for sedation drug. Balanced propofol sedation (BPS) refers to the administration of an opiate, a benzodiazepine, and propofol.
  Arms: balanced propofol group
Drug: propofol — propofol are used for sedation drug
  Arms: propofol alone group

SUMMARY:
Since introduction in 1989, propofol has gained wide acceptance for sedation during endoscopic procedures. The optimal sedation drug during esophagogastroendoscopy (EGD) is not established. Midazolam and propofol are used for sedation drug. Balanced propofol sedation (BPS) refers to the administration of an opiate, a benzodiazepine, and propofol. In this study, the investigators want to compare the patient satisfaction with EGD following balanced propofol sedation (BPS) versus propofol sedation alone.

ELIGIBILITY:
Inclusion Criteria:

1. over 19 years old, male and female
2. patients who have plan to get esophagogastroduodenoscopy (EGD)

Exclusion Criteria:

1. ASA class III or IV
2. Allergies to propofol, sulfites or eggs
3. patients who had surgery for esophagus, stomach or duodenum
4. inpatients
5. patients who had sleep apnea, gastroparesis or achalasia
6. patients who are taking sedative drugs more than 6 months
7. pregnancy
8. hypotension (systolic pressure less than 90mmHg), bradycardia (pulse rates less than 50 times per minute) or hypoxia (SpO2 less than 90%)
9. psychiatric or neurologic problems (ex. epilepsy or dementia)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-02-04 (Actual)

PRIMARY OUTCOMES:
visual analog scale | Within the 24 hours after EGD
  The patient satisfaction with EGD following balanced propofol sedation (BPS) versus propofol sedation alone

SECONDARY OUTCOMES:
complications rates | Within the 1 hour after EGD
  The recovery time after EGD following balanced propofol sedation versus propofol sedation alone. The safety after EGD following balanced propofol sedation versus propofol sedation alone

OTHER OUTCOMES:
complications rates | Within the 1 hour after EGD
  The safety after EGD following balanced propofol sedation versus propofol sedation alone
total dose of the sedation drugs | Within the 1 hour after EGD
  The economy after EGD following balanced propofol sedation versus propofol sedation alone
visual analog scale | Within the 1 hour after EGD
  The endoscopist's satisfaction with EGD following balanced propofol sedation (BPS) versus propofol sedation alone

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university College of Medicine, Seoul, Seoul, South Korea